CLINICAL TRIAL: NCT02137460
Title: Korean Brain Aging Study for Early Diagnosis and Prediction of Alzheimer's Disease
Acronym: KBASE
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Dong Young Lee, professor, Seoul National University Hospital
Other Study IDs: KBASE01; NRF-2013M3C7A1072998 (Other Grant/Funding Number: NRF-2013M3C7A1072998); NRF-2013M3C7A1069644 (Other Grant/Funding Number: NRF-2013M3C7A1069644); NRF-2014M3C7A1046042 (Other Grant/Funding Number: NRF-2014M3C7A1046042); NRF-2014M3C7A1046037 (Other Grant/Funding Number: NRF-2014M3C7A1046037)
Record Dates: First submitted 2014-05-08; First posted 2014-05-13 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Alzheimer's disease; Early diagnosis; Prediction; Biomarker; Imaging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, DNA, RNA, hair, and stool
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Young normal controls: * age : 20 ~ 55
  * without dementia, MCI, or other major neurological/psychiatric illness
- Elderly normal controls: * age : 55 ~ 90
  * without dementia, MCI, or other major neurological/psychiatric illness
- MCI (Mild cognitive impairment): * age : 55 ~ 90
  * without major neurological/psychiatric illness
  * concern regarding a change in cognition, lower performance in episodic memory domains that is greater than would be expected for the subject's age and educational background and preservation of independence in functional abilities
- AD (Alzheimer's diseases): * age: 55 ~ 90
  * National Institute of Aging and the Alzheimer's Association (NIA-AA) Probable AD dementia

SUMMARY:
This is a prospective cohort study for cognitively normal (young and old), mild cognitive impairment, and Alzheimer's disease people

DETAILED DESCRIPTION:
The aim of the study is 1) to search new biomarkers and develop clinically applicable early diagnosis and prediction methods of Alzheimer's disease, and 2) to investigate how the proposed lifetime risk and protective factors for Alzheimer's disease contribute to pathological hallmarks of AD or other brain changes in living human through annual comprehensive clinical and neuropsychological evaluation and biannual brain imaging (MRI and MRA, Fluorodeoxyglucose(FDG)-PET, Pittsburgh compound B (PiB)-PET), AV--1451 PET, and body specimen (blood, gene, and hair) analysis.

* Note: AV-1451 PET will not be applied to whole subjects, but to 210 subjects (30 young CN, 60 old CN, 60 MCI, and 60 AD).

ELIGIBILITY:
Participants will be classified as either Alzheimer's disease(AD) group, mild cognitive impairment(MCI) group, elderly normal controls or young normal controls. Specific inclusion criteria for each group is described below.

[Inclusion criteria: AD]

* Age : 55 - 90
* Clinical Dementia Rating (CDR)=0.5 or 1
* Diagnostic and Statistical Manual-IV(DSM-IV) criteria for dementia
* National Institute of Aging and the Alzheimer's Association (NIA-AA) Probable AD dementia
* Study partner or caregiver to accompany patient to all scheduled visits
* Written informed consent

[Inclusion criteria: MCI (amnestic)]

* Age : 55 - 90
* Clinical Dementia Rating (CDR)=0.5
* Concern regarding a change in cognition (obtained from the subject, from an informant who knows the subject, or from a skilled clinician observing the subject)
* Lower performance in episodic memory domains that is greater than would be expected for the subject's age and educational background
* Preservation of independence in functional abilities
* Study partner or caregiver to accompany subject to all scheduled visits
* Written informed consent

[Inclusion criteria: Elderly normal controls]

* Age : 55 - 90
* Clinical Dementia Rating (CDR)=0
* Those with contactable Informant
* Written informed consent

[Inclusion criteria: Young normal controls]

* Age : 20 - 55
* Clinical Dementia Rating (CDR)=0
* Written informed consent

[Exclusion criteria: general]

* Past history or presence of major psychiatric illness (e.g. schizophrenia, bipolar disorder, alcohol/substance abuse or dependence, delirium)
* Significant neurologic or medical condition that can influence the mental state
* Contraindications for MRI scan (e.g. pacemaker, claustrophobia)
* Illiteracy
* Significant visual or hearing difficulty
* Taking investigational drug
* In pregnancy or breast-feeding

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Young and elderly normal controls: community-based population AD and MCI: clinic or community-based population
Sampling Method: Non-Probability Sample
Enrollment: 721 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
The amount of brain amyloid deposition | baseline
  Group difference in baseline brain amyloid deposition (on PIB PET) and the relationship between the amount of brain amyloid deposition and clinical, neuropsychological, neuroimaging, genetic, biochemical measurement will be investigated.

SECONDARY OUTCOMES:
Group difference for each clinical, neuropsychological, structural and functional neuroimaging, tau imaging, genetic, biochemical measures | baseline
  Group difference for clinical, neuropsychological, structural and functional neuroimaging, tau imaging, genetic, biochemical variables and correlations among these variables will be investigated.
Change of brain amyloid deposition | baseline, 2yr, 4yr
  The change of brain amyloid deposition and its relation to the clinical, neuropsychological, neuroimaging, genetic and biochemical variables will be assessed.
Change of clinical, neuropsychological measures | baseline, 1yr, 2yr,3yr, 4yr
  The change of clinical, neuropsychological measurement and the relationship between these variables and other biomarkers will be assessed.
Change of structural and functional neuroimaging measures | baseline, 2yr, 4yr
  The change of structural and functional MRI measures and glucose metabolism of the brain the relationship between these variables and other clinical, neuropsychological, neuroimaging, biochemical, genetic biomarkers will be assessed.
Change of biochemical measures | baseline, 2yr, 4yr
  The change of blood or hair-based biochemical measures and the relationship between these variables and other clinical, neuropsychological, neuroimaging, biochemical, genetic biomarkers will be assessed.
Chage of tau imaging measures | 2yr, 4yr
  The change of tau PET imaging measures and the relationship between these measures and other clinical, neuropsychological, neuroimaging, biochemical, genetic biomarkers will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Young Lee, MD, PhD, Principal Investigator — Department of Psychiatry, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea